CLINICAL TRIAL: NCT00121537
Title: A Prospective Study to Determine the Utility of Vacuum Assisted Closure (VAC) Compared to Conventional Saline Dressing Changes With Regards to Lower Extremity Fasciotomy Wound Healing, Complications, Cost and Patient and Nursing Satisfaction
Brief Title: Study to Determine the Utility of Wound Vacuum Assisted Closure (VAC) Compared to Conventional Saline Dressing Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: terminated, due to lack enrollment,
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 045-1502-226
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Wounds; Compartment Syndromes
Keywords: wounds-open
MeSH Terms: conditions — Wounds and Injuries; Compartment Syndromes

INTERVENTIONS:
Device: Wound Care -Wound Vacuum Assisted Closure (VAC)
Procedure: Wound Care - Wet to Dry Dressing Changes

SUMMARY:
The purpose of this study is to look at the use of the wound vacuum assisted closure (VAC) versus standard wet to dry dressing in treating lower leg fasciotomies.

ELIGIBILITY:
Inclusion Criteria:

* four compartment fasciotomies performed on one or both lower extremities
* subject and/or subject's legally authorized representative (next-of-kin) has voluntarily signed and dated informed consent.

Exclusion Criteria:

* inability to place wound VAC
* contraindications for wound VAC use
* pregnant females
* prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Rate of wound healing

SECONDARY OUTCOMES:
Time to delayed primary wound closure
Time to completion of secondary healing
Patient satisfaction
Nurse satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: John G Myers, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States